CLINICAL TRIAL: NCT00030628
Title: A Phase III Randomized Trial Of The Role Of Whole Brain Radiation Therapy In Addition To Radiosurgery In The Management Of Patients With One To Three Cerebral Metastases
Brief Title: Radiosurgery With or Without Whole-Brain Radiation Therapy in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z0300; ACOSOG-Z0300; CDR0000069183 (Other: NCI Physician Data Query)
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- radiosurgery (Experimental): Patients undergo radiosurgery.
  Quality of life is assessed at baseline, the beginning of each treatment, at week 6, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 2 years.
  Interventions: Radiation: radiation therapy; Procedure: surgery
- radiosurgery + WBRT (Experimental): Patients undergo radiosurgery. Within 14 days, patients then undergo whole brain radiotherapy 5 days a week for 2.5 weeks.
  Quality of life is assessed at baseline, the beginning of each treatment, at week 6, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 2 years.
  Patients are followed at weeks 6 and 12, every 3 months for 9 months, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.
  Interventions: Radiation: radiation therapy; Procedure: surgery; Radiation: WBRT

INTERVENTIONS:
Radiation: radiation therapy
Procedure: surgery
Radiation: WBRT
  Arms: radiosurgery + WBRT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Radiosurgery may be able to deliver x-rays directly to the tumor and cause less damage to normal tissue. It is not yet known if radiosurgery is more effective with or without whole-brain radiation therapy in treating brain metastases.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiosurgery with or without whole-brain radiation therapy in treating patients who have brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with 1 to 3 cerebral metastases treated with radiosurgery with or without whole brain radiotherapy.
* Compare the time to CNS failure (brain) in patients treated with these regimens.
* Compare the quality of life, duration of functional independence, and long-term neurocognitive status in patients treated with these regimens.
* Compare the post-treatment toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (60 and over vs under 60), extracranial disease (controlled for more than 3 months vs controlled for 3 months or less), and number of brain metastases (1 vs more than 1). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiosurgery.
* Arm II: Patients undergo radiosurgery. Within 14 days, patients then undergo whole brain radiotherapy 5 days a week for 2.5 weeks.

Quality of life is assessed at baseline, the beginning of each treatment, at week 6, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 2 years.

Patients are followed at weeks 6 and 12, every 3 months for 9 months, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 480 patients (240 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral metastases meeting all of the following requirements:

  * 1-3 de novo lesions
  * Metastases must be from a histologically confirmed extracerebral primary site, another metastatic site, or from the metastatic brain lesion(s)
  * Each lesion must be less than 3.0 cm by contrasted MRI of the brain
  * Lesions must not be within 5 mm of optic chiasm or within the brainstem
* No primary germ cell tumor, small cell carcinoma, or lymphoma
* No leptomeningeal metastases
* Eligible for treatment with gamma knife or linear accelerator-based radiosurgery
* Performance status - ECOG 0-2
* Performance status - Zubrod 0-2
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Male patients must continue to use contraception for 3 months after the completion of radiotherapy
* No pacemaker or other MRI-incompatible metal in body
* No known allergy to gadolinium
* Deemed to be at low risk for recurrence from any prior malignancies
* At least 7 days since prior chemotherapy
* Concurrent hormonal agents allowed
* Concurrent steroids allowed
* No prior cranial radiotherapy
* No prior resection of cerebral metastasis
* Concurrent anticonvulsants allowed provided therapeutic serum/plasma level maintained before study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2001-12; Primary Completion 2005-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 6 months

SECONDARY OUTCOMES:
Time to CNS failure | Up to 4 years
Change in QOL between SRS and SRS + WBRT treatment groups using the FACT-BR questionnaire | From baseline to up to 3 months
Change in the duration of functional independence using the Barthel ADL Index score | From baseline to up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Asher, MD, FACS, Study Chair — Carolina Neurosurgery and Spine Associates
Locations (37):
- United States (37):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mount Diablo Regional Cancer Center, Concord, California
  - Sutter Cancer Center, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - John Muir Comprehensive Cancer Center at John Muir Medical Center, Walnut Creek, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - University of Illinois Medical Center, Chicago, Illinois
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - John F. Kennedy Medical Center, Edison, New Jersey
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - American College of Surgeons Oncology Group, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center - Shadyside Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Methodist Cancer Center at Methodist University Hospital, Memphis, Tennessee
  - American Fork Hospital, American Fork, Utah
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin